CLINICAL TRIAL: NCT02107417
Title: The Use of Transcutaneous Electrical Nerve Stimulation (Tens) in Reducing Symptoms of Peripheral Neuropathy Induced by Antineoplastic Chemotherapy
Brief Title: Study of TENS in Reducing Symptoms of Peripheral Neuropathy Induced by Chemotherapy
Acronym: CIPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Nacional de Cancer, Brazil (Other Government); Instituto do Cancer do Estado de São Paulo (Other); Hospital de Câncer de Barretos (Other); Centro de Estudos e Pesquisas Oncológicas (CEPO) (Unknown); Centro de Oncologia do Hospital Universitário São Francisco (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USP-2014-NPIQ
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Neuropathy; Pain; Paresthesia; Neuritis
Keywords: chemotherapy; pain; paresthesia; Physiotherapy; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain; Paresthesia; Neuritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (EG) - TENS active (Experimental): Experimental Group (EG) - TENS active: who will receive the application of active TENS. The participants of these group will receive TENS active within the following parameters: VF mode TENS with a variable frequency between 7 Hz and 65 Hz. It has a pulse width of 200 µs, this is the highest tolerable intensity while still remaining comfortable for the patient. It has an application time of 60 minutes with the highest tolerable intensity, while still remaining comfortable for the patient.
  Interventions: Device: active TENS
- Control Group (CG)- Placebo TENS (Sham Comparator): Control Group (CG) who will be administering the placebo TENS.The participants of these group will receive TENS within the following parameters: VF mode TENS with a variable frequency between 7 Hz and 65 Hz. It has a pulse width of 200 µs, . It has an application time of 60 minutes The TENS-placebo will be applied where no current will be emitted.
  Interventions: Device: placebo TENS

INTERVENTIONS:
Device: active TENS — Experimental Group (EG) who will receive the application of active TENS. The participants of these group will receive TENS within the following parameters: VF mode TENS with a variable frequency between 7 Hz and 65 Hz. It has a pulse width of 200 µs, this is the highest tolerable intensity while still remaining comfortable for the patient. It has an application time of 60 minutes with the highest tolerable intensity, while still remaining comfortable for the patient.
  Other Names: Experimental Group (EG)- active TENS
  Arms: Experimental Group (EG) - TENS active
Device: placebo TENS — who will be administering the placebo TENS.The participants of these group will receive TENS within the following parameters: VF mode TENS with a variable frequency between 7 Hz and 65 Hz. It has a pulse width of 200 µs, this is the highest tolerable intensity while still remaining comfortable for the patient. It has an application time of 60 minutes The TENS-placebo will be applied where no current will be emitted. Patients in the placebo group will only feel the tingling for 45 seconds and after this period the device will not emit impulses, but it will work for 1 hour.
  Arms: Control Group (CG)- Placebo TENS

SUMMARY:
This study aims to investigate the effects of Transcutaneous Electrical Nerve Stimulation (TENS) in reducing the symptoms of pain and numbness and improve the daily lives of cancer patients who have Chemotherapy-induced peripheral neuropathy (CIPN).

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) results from damage or dysfunction of the peripheral nerves and is one of the most common side effects of antineoplastic chemotherapy when neurotoxic drugs are used. Pain and paresthesia symptoms are prevalent, causing chronic discomfort and loss of functional abilities whilst also interfering negatively with quality of life and the patient's autonomy. In a pilot study of patients with CIPN, there was evidence that Transcutaneous Electrical Nerve Stimulation (TENS) improved the painful symptoms of patients with CIPN. This study aims to investigate the effects of TENS in reducing the symptoms of pain and numbness and improve the daily lives of cancer patients who have CIPN.

1. Primary Objectives Evaluate the effects of TENS in the reduction of symptoms related to peripheral neuropathy due to chemotherapy treatment of a high and moderate neurotoxic potential in cancer patients.

Secondary Objectives:

* Evaluate the therapeutic response of TENS with frequency variation (FV) in symptoms of paresthesia
* Evaluate the therapeutic response of TENS with frequency variation (FV) in activities of the daily lives of patients
* Evaluate the therapeutic response of TENS with frequency variation (FV) in symptoms of neuropathic pain.
* Evaluate the factors associated with better treatment response in paresthesia, in pain and activities of daily living.

Eligibility criteria: The participants of the research will include patients with any cancer diagnosis who are being subjected to chemotherapy in either adjuvant or neoadjuvant therapy, containing in its protocol at least one chemotherapeutic drug of moderate and high neurotoxic potential.

The participants of the research will receive TENS within the following parameters: VF mode TENS with a variable frequency between 7 Hz and 65 Hz. It has a pulse width of 200 µs, this is the highest tolerable intensity while still remaining comfortable for the patient. It has an application time of 60 minutes with the highest tolerable intensity, while still remaining comfortable for the patient. The treatment will be given on the same day as the chemotherapy, and will be given from home within 3 cycles. The participants will be divided into 2 groups: Experimental Group (EG) who will be administering the active TENS and the Control Group (CG) who will be administering the placebo TENS. The evaluation of the effects will be measured through the following instruments: Classification of neuropathy by the CTCAE (Common Terminology Criteria for Adverse Events) version 4.02 2009, scale of functionality ECOG, the Questionnaire of Neurotoxicity Induced by Antineoplastics (QNIA) for the evaluation of the symptoms of CIPN, and the Analogue Visual Scale (AVS) to assess the symptoms of pain and paresthesia. The error α is estimated at 5%.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who are being subjected to chemotherapeutic treatment with drugs or association of drugs with high and moderate neurotoxic degree and who present neuropathic pain and / or peripheral sensory neuropathy grade I and II of the CTCAE scale (Appendix A).
* Patients showing symptoms of peripheral neuropathy in the first cycle of chemotherapeutic treatment with three points on the visual analogue scale of pain and paresthesia.
* Patients aged between 18 and 70 years.
* Patients without Diabetes Mellitus before and during chemotherapy treatment.
* Patients who have not undergone previous chemotherapy regimens with neurotoxic drugs.
* Patients with ECOG performance status ≤ 2 (Karnofsky ≥ 50%).
* Patients that do not have a cardiac pacemaker.
* Patients without changes in sensitivity prior to chemotherapy.
* Patients without skin lesions at the site or around the site of application of the electrodes.
* Patients without cognitive and comprehension difficulties.
* Agree to participate in the study by signing the Free and Clarified Term of Consent- FCTC

Exclusion Criteria:

* Patients who have already undergone chemotherapy previously with drugs or have had association with neurotoxic drugs which have presented neuropathic pain and/or sensory peripheral neuropathy.
* Patients who have previously had acupuncture for the treatment of neuropathic pain and/or sensory peripheral neuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of TENS in the reduction of symptoms related to peripheral neuropathy due to chemotherapy treatment of a high and moderate neurotoxic potential in cancer patients. | At each chemotherapeutic cycle, for the duration of three cycles (approximately 9 weeks).

SECONDARY OUTCOMES:
Evaluate the therapeutic response of TENS in symptoms of paresthesia | At each chemotherapeutic cycle, for the duration of three cycles (approximately 9 weeks).
Evaluate the therapeutic response of TENS in activities of the daily lives of patients. | At each chemotherapeutic cycle, for the duration of three cycles (approximately 9 weeks).
Evaluate the therapeutic response of TENS in symptoms of neuropathic pain. | At each chemotherapeutic cycle, for the duration of three cycles (approximately 9 weeks).
Evaluate the factors associated with better treatment response in paresthesia, in pain and activities of daily living. | At each chemotherapeutic cycle, for the duration of three cycles (approximately 9 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Tania Tonezzer, B.S, Principal Investigator — Post-Graduation Student of Rehabilitation Science Program from Department of Speech Therapy, Physical Therapy and Occupational Therapy, São Paulo University, São Paulo, Brazil.
Locations (1):
- Instituto do Câncer de São Paulo, São Paulo, São Paulo, Brazil